CLINICAL TRIAL: NCT04284670
Title: The Effect of Eccentric Training on Anthropometrics, Physical Fitness and Bone Strength in Overweight Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, Dan Nemet, MD, Director, Child Health and Sports Center, Meir Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: MeirMc0163-19CTIL
Record Dates: First submitted 2019-09-25; First posted 2020-02-26 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Childhood Obesity
Keywords: eccentric training; childhood obesity; decline treadmill
MeSH Terms: conditions — Pediatric Obesity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Eccentric treadmill training (Experimental): The intervention group will perform an 8 week program, 2 sessions a week for a total of 16 sessions. training will be done on a designated negative gradient treadmill. first two session will be in -5% gradient. sessions 3,4 and 5 will be in -10% gradient, all of the following sessions will be in -15% gradient. exercise intensity will be 70%-80% out of maximal heart-rate. Session length will gradually increase by one minute each training, starting from 10 minutes at the first session, up to 25 minutes on final sessions. each training will start and end with a 2 minutes of warm up and calm down under neutral gradient. Every two minutes of training, Visual Analog Scale and Rating of Perceived Exertion data will be collected from the participants.
  Interventions: Other: EXERCISE
- Control group (Experimental): The control group will receive the same amount of training under neutral gradient surface(0%).The program will be 8 weeks while in each week there will be two exercise sessions and a total of 16 sessions. Session length will gradually increase by one minute each training, starting from 10 minutes at the first session, up to 25 minutes on final sessions. Training intensity will be 70%-80% out of maximal heart-rate.
  Interventions: Other: EXERCISE

INTERVENTIONS:
Other: EXERCISE — The intervention group will perform an 8 week program, 2 sessions a weak for a total of 16 sessions. training will be done on a designated negative gradient treadmill, first two session will be in -5% gradient. sessions 3,4 and 5 will be in -10% gradient, all of the following sessions will be in -15% gradient. exercise intensity will be 70%-80% out of maximal heart-rate. Session length will gradually increase by one minute each training, starting from 10 minutes at the first session, up to 25 minutes on final sessions. each training will start and end with a 2 minutes of warm up and calm down under neutral gradient. Every two minutes of training, Visual Analog Scale and Rating of Perceived Exertion data will be collected from the participants.

SUMMARY:
The purpose of this study is to examine the effects of aerobic eccentric training in overweight and obese children.

DETAILED DESCRIPTION:
recent studies have shown that similarly to regular exercise, aerobic ECcentric Contraction (ECC) exercise induces changes in the musculoskeletal system while using lower energy consumption, due to the fact that eccentric training creates greater force in the muscle.

most of the studies in this subject were done on healthy or overweight adults. therefore, the effect of aerobic eccentric training on children is still unknown. this study wants to test the impact of eccentric training on overweight and obese children.

this study will include approximately 100 overweight and obese children (boys and girls), aged 5-18 years. participants will be recruited from the population of overweight children from children sports medical center 'Meir' in Kfar Saba, Israel. participants will be randomly divided into two groups (intervention and control). Participants and their parents will sign a consent form before entering the study.

Each participant will undergo a series of tests including: anthropometrics (height, weight, bmi, body composition by BIA), fitness tests (Maximal distance achieved in a 12min outdoor run\walk, Vertical jump, Standing long jump, 4X10 meter sprint run), quadriceps and hamstrings strength test (hand-held dynamometer MicroFet2), bone strength (bone sonometer), ankle and tibial kinematic(accelerometers+ video of foot strike).

Intervention group will then perform an 8 week (16 sessions) ECC training program on a decline treadmill, the program will include two weeks of habituation to lower as possible DOMS (delayed onset muscle soreness) and possible injuries, training length and intensity will be gradually increasing over the time of the program, maximal negative gradient will be -15% at the end of the program.

Control group will perform the same amount of training (volume, intensity and frequency) on a neutral gradient surface. After completing the training program each participant will perform again the series of tests. Once all the data is collected, statistical test will be performed in order to learn about the effect of ECC training program on overweight and obese children.

ELIGIBILITY:
Inclusion Criteria:

* Children and adolescents aged 5-18.
* Children and adolescents with overweight defined as BMI percentile over 85%.
* Children and adolescents who are able to perform moderate physical activity.
* Children and adolescents that participate in 'Meir' hospital sports and health centre.

Exclusion Criteria:

* Participant that does not wish to participate - will not be obligated to do so, and shall not participate in the study.
* Participants with orthopaedic history in the past two years.

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-07-01 (Estimated); Study Completion 2021-11-01 (Estimated)

PRIMARY OUTCOMES:
Physical fitness | 8 weeks
  participants will show changes in physical activity-run/walk perseverance time.
BMI Percentile | 8 weeks
  participants will show changes in BMI Percentile
Muscle strength by Hand-held Dynamometer(newton) | 8 weeks
  participants will show changes in quadriceps and hamstring group muscles strength.
Tibial Bone Strength by US(m/s) | 8 weeks
  participants will show changes in tibial bone strength
Peak Positive Acceleration (PPA) | 8 weeks
  participants will show changes in tibial bone acceleration.

CONTACTS AND LOCATIONS:
Locations (1):
- 'Meir children's sport and health center', Kfar Saba, Israel